CLINICAL TRIAL: NCT03858426
Title: Prospective Multicenter Nationwide Registry of Children With Eosinophilic Esophagitis
Acronym: RENESE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Espanola de Gastroenterologia, Hepatologia y Nutricion Pediatrica (Other)
Responsible Party: Principal Investigator, Carolina Gutierrez Junquera, Principal Investigator, Sociedad Espanola de Gastroenterologia, Hepatologia y Nutricion Pediatrica
Other Study IDs: RENESE
Record Dates: First submitted 2018-10-11; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; PPIs, children, elimination diet, topical steroids
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with eosinophilic esophagitis: Inclusion criteria:
  * Children from 1 month to 18 years with a new diagnosis of eosinophilic esophagitis according to recent European guidelines (symptoms of esophageal dysfunction + eosinophilic infiltrate of the esophagus > 15 eos / CGA)
  * And they need to start treatment with one of the following options: PPI, diet excluding cow's milk and gluten, or swallowed corticosteroids
  Exclusion criteria:
  * Presence of pathological eosinophilia at the gastric or duodenal level (eosinophilic gastroenteritis)
  * Simultaneous treatment with more than one treatment modality (PPI, empirical elimination diet, swallowed corticosteroids).
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
1. Registry of demographic, clinical, endoscopic and histological data at baseline.
2. Registry of patients treated with PPI:

   * Clinical, endoscopic and histological response at 8-12 weeks of induction treatment
   * Clinical, endoscopic and histological response at 6 and 12 months weeks of maintenance treatment
3. Registry of patients treated with two foods elimination diet:

   * Clinical, endoscopic and histological response at 8-12 weeks of induction treatment
   * Identification of food trigger: milk, gluten or milk and gluten
   * Clinical, endoscopic and histological response at one year elimination of food trigger
   * Registry of adverse events
4. Registry of patients treated with swallowed steroids (budesonide or fluticasone):

   * Clinical, endoscopic and histological response at 8-12 weeks of induction treatment
   * Clinical, endoscopic and histological response at 6 months of maintenance steroid treatment
   * Registry of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Children from 1 month to 18 years with a new diagnosis of eosinophilic esophagitis (EoE) according to the recent European guidelines (symptoms of esophageal dysfunction + eosinophilic infiltrate of the esophagus > 15 eos / CGA)
* And that they need to start treatment with any of the following options: PPI, diet excluding cow's milk and gluten, or swallowed corticosteroids .

Exclusion Criteria:

* Presence of pathological eosinophilia at the gastric or duodenal level (eosinophilic gastroenteritis)
* Simultaneous treatment with more than one treatment modality (PPI, empirical elimination diet, swallowed corticosteroids).

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children from 1 month to 18 years with a new diagnosis of eosinophilic esophagitis according to the recent European guidelines
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Complete histological remission | 12 weeks
  Complete histological remission response defined as ≤5 eosinophils/hpf in all biopsies performed

SECONDARY OUTCOMES:
Partial histological remission | 12 weeks
  Partial histological remission response defined as 5-15 eosinophils /hpf in all biopsies
Clinical remission | 12 weeks
  Clinical remission (specific questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Puerta de Hierro Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided